CLINICAL TRIAL: NCT00530348
Title: A Phase 3 Randomized, Rater-Blinded Study Comparing Two Annual Cycles of Intravenous Alemtuzumab to Three-Times Weekly Subcutaneous Interferon Beta-1a (Rebif®) in Treatment-Naïve Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Comparison of Alemtuzumab and Rebif® Efficacy in Multiple Sclerosis, Study One
Acronym: CARE-MS I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAMMS323; ISRCTN21534255 (Registry Identifier: ISRCTN); ACTRN12608000435381 (Registry Identifier: ANZCTR); CARE-MS I (Other: NMSS); 2007-001161-14 (EudraCT Number)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Alemtuzumab; Interferon beta-1a

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alemtuzumab (Experimental)
  Interventions: Biological: Alemtuzumab
- Interferon Beta-1a (Active Comparator)
  Interventions: Biological: Interferon beta-1a

INTERVENTIONS:
Biological: Alemtuzumab — Alemtuzumab 12 milligram (mg) per day intravenous (IV) infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
  Other Names: Lemtrada
  Arms: Alemtuzumab
Biological: Interferon beta-1a — Interferon beta-1a 44 microgram (mcg) subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
  Other Names: Rebif®
  Arms: Interferon Beta-1a

SUMMARY:
The purpose of this study was to establish the efficacy and safety of alemtuzumab (Lemtrada™) as a treatment for relapsing-remitting multiple sclerosis (MS), in comparison with subcutaneous (SC) interferon beta-1a (Rebif®). The study had enrolled participants who had not previously received MS disease-modifying therapies. Participants had monthly laboratory tests and comprehensive testing every 3 months.

DETAILED DESCRIPTION:
Every participant had received active treatment; there was no placebo. Participants who qualified were randomly assigned to treatment with either alemtuzumab or SC interferon beta-1a at a 2:1 ratio (that is, 2 given alemtuzumab for every 1 given interferon beta-1a). Alemtuzumab was administered in two annual courses, once at the beginning of the study and again 1 year later. Interferon beta-1a was self-injected 3 times per week for 2 years. All participants were required to return to their study site every 3 months for neurologic assessment. In addition, safety-related laboratory tests were performed at least monthly. Participation in this study ended 2 years after the start of treatment for each participant. Additionally, participants who received alemtuzumab might be followed in CAMMS03409 (NCT00930553) an extension study for safety and efficacy assessments. Participants who received interferon beta-1a and completed 2 years on study might be eligible to receive alemtuzumab on the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Given written/signed informed consent
* Age 18 to 50 years old (inclusive) as of the date the informed consent form (ICF) was signed
* Diagnosis of MS per updated McDonald criteria, and cranial magnetic resonance imaging (MRI) scan demonstrating white matter lesions attributable to MS within 5 years of screening
* Onset of MS symptoms (as determined by a neurologist, either at screening or retrospectively) within 5 years of the date the ICF was signed
* Expanded Disability Status Scale (EDSS) score 0.0 to 3.0 (inclusive) at screening
* Greater than or equal to (>=) 2 MS attacks (first episode or relapse) occurring in the 24 months prior to the date the ICF was signed, with >=1 attack in the 12 months prior to the date the ICF was signed, with objective neurological signs confirmed by a physician, nurse practitioner, or other Genzyme-approved health-care provider and the objective signs could be identified retrospectively

Exclusion Criteria:

* Received prior therapy for MS other than corticosteroids, for example, alemtuzumab, interferons, intravenous immunoglobulin, glatiramer acetate, natalizumab, and mitoxantrone
* Exposure to azathioprine, cladribine, cyclophosphamide, cyclosporine A, methotrexate, or any other immunosuppressive agent other than systemic corticosteroid treatment
* Any progressive form of MS
* History of malignancy (except basal skin cell carcinoma)
* CD4 + , CD8 + count, B cell, or absolute neutrophil count less than (<) lower limit of normal (LLN) at screening
* Known bleeding disorder (for example, dysfibrinogenemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation, fibrinogen deficiency, or clotting factor deficiency)
* Significant autoimmune disease including but not limited to immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis
* Presence of anti-thyroid stimulating hormone (TSH) receptor (TSHR) antibodies (that is, above the LLN)
* Active infection or at high risk for infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 581 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (101):
- United States (36):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - Barrow Neurological Institute, St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Neurological Associates, Pompano Beach, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Idaho Falls Multiple Sclerosis Center, PLLC, Idaho Falls, Idaho
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerican Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Health Sciences Center, MS Specialty Clinic, Albuquerque, New Mexico
  - Empire Neurology, Latham, New York
  - Comprehensive Multiple Sclerosis Care Center at South Shore Neurologic Associates, P.C., Patchogue, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Medical Center (CMC), Neurosciences & Spine Institute (NSSI), Charlotte, North Carolina
  - The Ohio State University Medical Center, Multiple Sclerosis Center, Columbus, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - MS Center of Oklahoma, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital Neurosciences and Pain Research, Allentown, Pennsylvania
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Biomedical Research Alliance of NY, LLC, Franklin, Tennessee
  - Hope Neurology PC, Knoxville, Tennessee
  - Baylor College of Medicine, Maxine Mesinger MS Clinic, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
- DIABAID, Buenos Aires, Argentina
- Australia (9):
  - The Wesley Research Institute, Auchenflower, Queensland
  - Griffith University School of Medicine, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Department of Neurology, Ward 4 East, Parkville, Victoria
  - Concord Repatriation General Hospital, Concord
  - Westmead Hospital, Westmead
- Brazil (3):
  - Hospital da Restauracao, Av Governador Agamenon Magalhaes, Recife, Pernambuco
  - Hospital Sao Lucas PUC-RS, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas USP, São Paulo, São Paulo
- Canada (5):
  - University of Calgary and Foothills Medical Cenre, Calgary, Alberta
  - UBC Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Clinique Nuero-outaouais, Gatineau, Quebec
  - Clinique Neuro rive-sud, Recherche Sepmus, Inc., Greenfield Park, Quebec
- Croatia (5):
  - Clinical Hospital Centre Rijeka, Rijeka
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Centre "Sestre Milosrdnice", Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
  - General Hospital "Sveti Duh", Zagreb
- Czechia (2):
  - Department of Neurology, 1st Faculty of Medicine and General Teaching Hospital, Prague
  - Krajska zdravotni a.s., Hospital Teplice, Teplice
- Hopital Purpan, Toulouse, France
- Germany (6):
  - Judisches Krankenhaus Berlin, Berlin
  - Universitätsklinik Carl Gustav Carus Dresden, Dresden
  - Klinikum der Goethe Universität Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Oberhavelkliniken Hennigsdorf, Hennigsdorf
  - Asklepios Klinikum Brandenburg, Teupitz
- Mexico (2):
  - Hospital Angeles del Pedregal, Camino de Santa Teresa, Mexico City
  - Hospital Medica Sur CIF-BIOTEC, Mexico City
- Poland (4):
  - Clinical Neurology Centre Sp. z o.o. (Ltd), Krakow
  - Independent Public Healthcare Facility, Norbert Barlicki University Hospital No. 1 of the Medical University of Lodz, Lodz
  - Independent Public Teaching Hospital No. 4 in Lublin, Lublin
  - Heliodor Swiecicki Teaching Hospital of the Poznan University of Medical Sciences, Poznan
- Russia (12):
  - Research Medical Complex "Your Health" Ltd, Kazan'
  - Moscow City Hospital #11, Moscow
  - Moscow State Medical Institution City Clinical Hospital #11, Moscow
  - Scientific Neurology Center RAMS, Moscow
  - Municipal City Hospital #33, Nizhny Novgorod
  - Federal State Institution Siberian Rettitorial Medical Center under Federal Medical-Biological Agency of Russia, Novosibirsk
  - City Clinical Hospital #2, Pyatigorsk
  - Institute of Human Brain RAS, Saint Petersburg
  - Nikolaevskaya Hospital, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Samara Regional Clinical Hospital n.a. Kalinin, Samara
  - State Medical Institution: Republican Clinical Hospital n.a. G.G. Kuvatov, Ufa
- Serbia (5):
  - Clinical Centre Serbia, Institute for Neurology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical centre Kragujevac, Kragujevac
  - Clinical Center Nis, Clinic for neurology, Niš
  - Clinical Centre of Vojvodina, Clinic for neurology, Novi Sad
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Ukraine (5):
  - Chernihiv Regional Hospital, Chernihiv
  - Institute of Neurology, Psychiatry and Narcology under the Academy of Medical Sciences of Ukraine, Department of Neuroinfection and Multiple Sclerosis, Kharkiv
  - Hospoital of the Directorate of the Medical Corps within the Ukrainian Security Service, Neurology Department, Kyiv
  - Kyiv Municipal Clinical Hospital #4, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
- United Kingdom (4):
  - Department Of Neurosciences, Addenbrookes Hospital, Cambridge, England
  - Centre for Neuroscience & Trauma, Blizard Institute of Cell and Molecular Science, Barts and The London School of Medicine and Dentistry, London, England
  - University Hospital of Wales, Cardiff, Wales
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] Cohen JA, Coles AJ, Arnold DL, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Fisher E, Brinar VV, Giovannoni G, Stojanovic M, Ertik BI, Lake SL, Margolin DH, Panzara MA, Compston DA; CARE-MS I investigators. Alemtuzumab versus interferon beta 1a as first-line treatment for patients with relapsing-remitting multiple sclerosis: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1819-28. doi: 10.1016/S0140-6736(12)61769-3. Epub 2012 Nov 1. PMID 23122652
- [Derived] Ziemssen T, Bass AD, Van Wijmeersch B, Eichau S, Richter S, Hoffmann F, Armstrong NM, Chirieac M, Cunha-Santos J, Singer BA. Long-term efficacy and safety of alemtuzumab in participants with highly active MS: TOPAZ clinical trial and interim analysis of TREAT-MS real-world study. Ther Adv Neurol Disord. 2025 Feb 10;18:17562864241306575. doi: 10.1177/17562864241306575. eCollection 2025. PMID 39935588
- [Derived] Coles AJ, Achiron A, Traboulsee A, Singer BA, Pozzilli C, Oreja-Guevara C, Giovannoni G, Comi G, Freedman MS, Ziemssen T, Shiota D, Rawlings AM, Wong AT, Chirieac M, Montalban X. Safety and efficacy with alemtuzumab over 13 years in relapsing-remitting multiple sclerosis: final results from the open-label TOPAZ study. Ther Adv Neurol Disord. 2023 Sep 21;16:17562864231194823. doi: 10.1177/17562864231194823. eCollection 2023. PMID 37745914
- [Derived] Riera R, Torloni MR, Martimbianco ALC, Pacheco RL. Alemtuzumab for multiple sclerosis. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD011203. doi: 10.1002/14651858.CD011203.pub3. PMID 37272540
- [Derived] Dayan CM, Lecumberri B, Muller I, Ganesananthan S, Hunter SF, Selmaj KW, Hartung HP, Havrdova EK, LaGanke CC, Ziemssen T, Van Wijmeersch B, Meuth SG, Margolin DH, Poole EM, Baker DP, Senior PA. Endocrine and multiple sclerosis outcomes in patients with autoimmune thyroid events in the alemtuzumab CARE-MS studies. Mult Scler J Exp Transl Clin. 2023 Jan 3;9(1):20552173221142741. doi: 10.1177/20552173221142741. eCollection 2023 Jan-Mar. PMID 36619856
- [Derived] Coles AJ, Jones JL, Vermersch P, Traboulsee A, Bass AD, Boster A, Chan A, Comi G, Fernandez O, Giovannoni G, Kubala Havrdova E, LaGanke C, Montalban X, Oreja-Guevara C, Piehl F, Wiendl H, Ziemssen T. Autoimmunity and long-term safety and efficacy of alemtuzumab for multiple sclerosis: Benefit/risk following review of trial and post-marketing data. Mult Scler. 2022 Apr;28(5):842-846. doi: 10.1177/13524585211061335. Epub 2021 Dec 9. PMID 34882037
- [Derived] Kuhle J, Daizadeh N, Benkert P, Maceski A, Barro C, Michalak Z, Sormani MP, Godin J, Shankara S, Samad TA, Jacobs A, Chung L, Rӧsch N, Kaiser C, Mitchell CP, Leppert D, Havari E, Kappos L. Sustained reduction of serum neurofilament light chain over 7 years by alemtuzumab in early relapsing-remitting MS. Mult Scler. 2022 Apr;28(4):573-582. doi: 10.1177/13524585211032348. Epub 2021 Aug 11. PMID 34378446
- [Derived] Coles AJ, Arnold DL, Bass AD, Boster AL, Compston DAS, Fernandez O, Havrdova EK, Nakamura K, Traboulsee A, Ziemssen T, Jacobs A, Margolin DH, Huang X, Daizadeh N, Chirieac MC, Selmaj KW. Efficacy and safety of alemtuzumab over 6 years: final results of the 4-year CARE-MS extension trial. Ther Adv Neurol Disord. 2021 Apr 23;14:1756286420982134. doi: 10.1177/1756286420982134. eCollection 2021. PMID 34035833
- [Derived] Horakova D, Boster A, Bertolotto A, Freedman MS, Firmino I, Cavalier SJ, Jacobs AK, Thangavelu K, Daizadeh N, Poole EM, Baker DP, Margolin DH, Ziemssen T; CARE-MS I, CARE-MS II, and CAMMS03409 Investigators. Proportion of alemtuzumab-treated patients converting from relapsing-remitting multiple sclerosis to secondary progressive multiple sclerosis over 6 years. Mult Scler J Exp Transl Clin. 2020 Dec 18;6(4):2055217320972137. doi: 10.1177/2055217320972137. eCollection 2020 Oct-Dec. PMID 33414927
- [Derived] Ziemssen T, Bass AD, Berkovich R, Comi G, Eichau S, Hobart J, Hunter SF, LaGanke C, Limmroth V, Pelletier D, Pozzilli C, Schippling S, Sousa L, Traboulsee A, Uitdehaag BMJ, Van Wijmeersch B, Choudhry Z, Daizadeh N, Singer BA; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Efficacy and Safety of Alemtuzumab Through 9 Years of Follow-up in Patients with Highly Active Disease: Post Hoc Analysis of CARE-MS I and II Patients in the TOPAZ Extension Study. CNS Drugs. 2020 Sep;34(9):973-988. doi: 10.1007/s40263-020-00749-x. PMID 32710396
- [Derived] Comi G, Alroughani R, Boster AL, Bass AD, Berkovich R, Fernandez O, Kim HJ, Limmroth V, Lycke J, Macdonell RA, Sharrack B, Singer BA, Vermersch P, Wiendl H, Ziemssen T, Jacobs A, Daizadeh N, Rodriguez CE, Traboulsee A; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy of alemtuzumab in relapsing-remitting MS patients who received additional courses after the initial two courses: Pooled analysis of the CARE-MS, extension, and TOPAZ studies. Mult Scler. 2020 Dec;26(14):1866-1876. doi: 10.1177/1352458519888610. Epub 2019 Nov 25. PMID 31762387
- [Derived] Van Wijmeersch B, Singer BA, Boster A, Broadley S, Fernandez O, Freedman MS, Izquierdo G, Lycke J, Pozzilli C, Sharrack B, Steingo B, Wiendl H, Wray S, Ziemssen T, Chung L, Margolin DH, Thangavelu K, Vermersch P. Efficacy of alemtuzumab over 6 years in relapsing-remitting multiple sclerosis patients who relapsed between courses 1 and 2: Post hoc analysis of the CARE-MS studies. Mult Scler. 2020 Nov;26(13):1719-1728. doi: 10.1177/1352458519881759. Epub 2019 Nov 1. PMID 31675266
- [Derived] Okai AF, Amezcua L, Berkovich RR, Chinea AR, Edwards KR, Steingo B, Walker A, Jacobs AK, Daizadeh N, Williams MJ; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy and Safety of Alemtuzumab in Patients of African Descent with Relapsing-Remitting Multiple Sclerosis: 8-Year Follow-up of CARE-MS I and II (TOPAZ Study). Neurol Ther. 2019 Dec;8(2):367-381. doi: 10.1007/s40120-019-00159-2. Epub 2019 Oct 25. PMID 31654272
- [Derived] Li Z, Richards S, Surks HK, Jacobs A, Panzara MA. Clinical pharmacology of alemtuzumab, an anti-CD52 immunomodulator, in multiple sclerosis. Clin Exp Immunol. 2018 Dec;194(3):295-314. doi: 10.1111/cei.13208. Epub 2018 Oct 1. PMID 30144037
- [Derived] Havrdova E, Arnold DL, Cohen JA, Hartung HP, Fox EJ, Giovannoni G, Schippling S, Selmaj KW, Traboulsee A, Compston DAS, Margolin DH, Thangavelu K, Rodriguez CE, Jody D, Hogan RJ, Xenopoulos P, Panzara MA, Coles AJ; CARE-MS I and CAMMS03409 Investigators. Alemtuzumab CARE-MS I 5-year follow-up: Durable efficacy in the absence of continuous MS therapy. Neurology. 2017 Sep 12;89(11):1107-1116. doi: 10.1212/WNL.0000000000004313. Epub 2017 Aug 23. PMID 28835401
- [Derived] Arnold DL, Fisher E, Brinar VV, Cohen JA, Coles AJ, Giovannoni G, Hartung HP, Havrdova E, Selmaj KW, Stojanovic M, Weiner HL, Lake SL, Margolin DH, Thomas DR, Panzara MA, Compston DA; CARE-MS I and CARE-MS II Investigators. Superior MRI outcomes with alemtuzumab compared with subcutaneous interferon beta-1a in MS. Neurology. 2016 Oct 4;87(14):1464-1472. doi: 10.1212/WNL.0000000000003169. Epub 2016 Sep 2. PMID 27590291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 101 investigational sites in Argentina, Australia, Brazil, Canada, Croatia, the Czech Republic, France, Germany, Mexico, Poland, Russia, Serbia, Sweden, Ukraine, the United Kingdom (UK), and the United States (US) between August 28, 2007 and April 27, 2011.
Groups:
- Interferon Beta-1a: Interferon beta-1a (Rebif®) 44 microgram (mcg) subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
- Alemtuzumab: Alemtuzumab (Lemtrada™) 12 milligram (mg) per day intravenous (IV) infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
Period: Overall Study
Arm/Group | Interferon Beta-1a | Alemtuzumab
Started | 195 (Randomized.) | 386 (Randomized.)
Treated | 187 (All randomized participants who received at least 1 dose of study drug.) | 376 (All randomized participants who received at least 1 dose of study drug.)
Completed | 173 | 367
Not Completed | 22 | 19
Not completed — Adverse Event | 5 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Randomised in error | 1 | 0
Not completed — Noncompliance with inclusion criterion 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Interferon Beta-1a: Interferon beta-1a 44 mcg subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
- Alemtuzumab: Alemtuzumab 12 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Alemtuzumab | Total
Number analyzed (Participants) | 187 | 376 | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.48) | 33.0 (8.03) | 33.1 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 243 | 365
  Male | 65 | 133 | 198
Time Since First Relapse [Mean (Standard Deviation); unit: years] | 2.0 (1.32) | 2.1 (1.36) | 2.1 (1.35)
Number of Relapse Episodes in the Preceding 2 Years [Number; unit: participants] — Number of participants with 1, 2 or greater than or equal to 3 relapses are reported.
  participants
    1 Relapse | 3 | 12 | 15
    2 Relapses | 118 | 215 | 333
    Greater than or equal to 3 Relapses | 66 | 149 | 215
Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that quantifies disability in participants with multiple sclerosis (MS). It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  units on a scale | 2.0 (0.79) | 2.0 (0.81) | 2.0 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Accumulation of Disability (SAD)
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score: 0 (normal neurological examination) to 10 (death due to MS). As measured by EDSS score, SAD was defined as increase of at least 1.5 points for participants with Baseline score of 0 and increase of at least 1.0 point for participants with a Baseline score of 1.0 or more; and the increase persisted for at least next 2 scheduled assessments, that is, 6 consecutive months. Onset date of SAD was date of first EDSS assessment that began 6 month consecutive period of SAD. Participants who did not reach SAD endpoint were censored at their last visit. Percentage of participants with SAD, estimated by Kaplan-Meier (KM) method, was reported.
Time Frame: Up to 2 years
Population: FAS population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants with SAD
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 187 | 376
percentage of participants with SAD | 11.12 [7.32 to 16.71] | 8.00 [5.66 to 11.24]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; Cox proportional hazards (PH) regression model with robust variance estimation using treatment group and geographic region as covariates was used; Test type: Superiority or Other; p = 0.2173, Cox Proportional Hazards Regression — Hochberg method was used to adjust for the two co-primary outcomes; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.40 to 1.23]

2. Primary Outcome: Annualized Relapse Rate
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to multiple sclerosis that lasted for at least 48 hours, that were present at normal body temperature, and that were preceded by at least 30 days of clinical stability. Annualized relapse rate was estimated through negative binomial regression with robust variance estimation and covariate adjustment for geographic region using observed number of relapses as dependent variable, the log total amount of follow-up from date of first study treatment for each participant as an offset variable, and treatment group and geographic region as model covariates.
Time Frame: Up to 2 years
Population: FAS population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 187 | 376
relapses per participant per year | 0.39 [0.29 to 0.53] | 0.18 [0.13 to 0.23]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; Proportional means regression model with robust variance estimation and covariate adjustment for geographic region was used; Test type: Superiority or Other; p < 0.0001, Proportional means regression — Hochberg method was used to adjust for the two co-primary outcomes; Rate ratio = 0.45, 95% CI 2-sided [0.32 to 0.63]

3. Secondary Outcome: Percentage of Participants Who Were Relapse Free at Year 2
Description: Participants were considered relapse free at Year 2 if they did not experience a relapse from the date of first study treatment to study completion at 24 months. Percentage of participants who were relapse free at Year 2, estimated using the KM method, was reported.
Time Frame: Year 2
Population: FAS population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 187 | 376
percentage of participants | 58.69 [51.12 to 65.50] | 77.59 [72.87 to 81.60]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; Cox PH regression model with robust variance estimation, covariate adjustment for geographic region, was used. Secondary endpoints were analyzed sequentially as: Proportion of participants relapse free at Year 2, Change from baseline in EDSS, Percent change from Baseline in magnetic resonance imaging-T2 hyperintense lesion volume at Year 2, Acquisition of disability measured by multiple sclerosis functional composite. Each endpoint could only be formally tested if prior endpoint was significant; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Regression; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.33 to 0.61]

4. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Year 2
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS). Change was calculated by subtracting Baseline value from value at Year 2.
Time Frame: Baseline, Year 2
Population: FAS population included all randomized participants who received at least 1 dose of study drug. Here, number of participants analyzed was subset of FAS who had EDSS assessment at both Baseline and end-of-study (Year 2).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 173 | 366
units on a scale | -0.2 (1.05) [-0.29 to 0.01] | -0.2 (0.87) [-0.25 to -0.02]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; The analysis was performed using Wei-Lachin method for non-parametric analysis of repeated measures. Secondary endpoints were analyzed sequentially as: Proportion of participants relapse free at Year 2, Change from baseline in EDSS, Percent change from Baseline in magnetic resonance imaging-T2 hyperintense lesion volume at Year 2, Acquisition of disability measured by multiple sclerosis functional composite. Each endpoint could only be formally tested if prior endpoint was significant; Test type: Superiority or Other; p = 0.4188, Wei-Lachin

5. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score at Year 2
Description: MSFC is a multidimensional measure consisting of quantitative tests of ambulation (Timed 25-Foot Walk), manual dexterity (9-Hole Peg Test; 9HPT), and cognitive function (Paced Auditory Serial Addition Test; PASAT). The MSFC score was calculated as the mean of the Z-scores of the 3 components. A Z-score was calculated by subtracting the mean of the reference population from the test result, then dividing by the standard deviation of the reference population. Higher Z-scores reflected better neurological function and a positive change from Baseline indicates improvement. An increase in score indicated an improvement (Z-score range: -3 to +3). Acquisition of disability was measured by change from Baseline in MSFC score at Year 2.
Time Frame: Baseline, Year 2
Population: FAS population included all randomized participants who received at least 1 dose of study drug. Here, number of participants analyzed signifies subset of FAS who had MSFC score assessment at Baseline; 'n' signifies participants who had MSFC score assessment at Baseline (for Baseline) and at both Baseline and Year 2 (for change at Year 2).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 186 | 375
Z-score
  Baseline (n=186, 375) | 0.05 (0.629) | -0.02 (0.695)
  Change at Year 2 (n=172, 362) | 0.07 (0.450) | 0.15 (0.516)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; Change at Year 2: analysis was performed using Wei-Lachin method for non-parametric analysis of repeated measures. Secondary endpoints were analyzed sequentially as: Proportion of participants relapse free at Year 2, Change from baseline in EDSS, Percent change from Baseline in magnetic resonance imaging-T2 hyperintense lesion volume at Year 2, Acquisition of disability measured by MSFC. Each endpoint could only be formally tested if prior endpoint was significant; Test type: Superiority or Other; p = 0.0115, Wei-Lachin

6. Secondary Outcome: Percent Change From Baseline in Magnetic Resonance Imaging Time Constant 2 (MRI-T2) Hyperintense Lesion Volume at Year 2
Description: Percent change in MS lesion volume as measured by MRI-T2 scan was calculated from MRI-T2-weighted scans as the following: (lesion volume at 2 years - lesion volume at Baseline)*100/ (lesion volume at Baseline).
Time Frame: Baseline, Year 2
Population: FAS population included all randomized participants who received at least 1 dose of study drug. Here, number of participants analyzed was subset of FAS who had assessment for T2 volume at both Baseline and end-of-study (Year 2).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Interferon Beta-1a | Alemtuzumab
Number analyzed (Participants) | 177 | 364
percent change | -6.68 (32.44) [-20.7 to 2.5] | -10.28 (22.58) [-19.6 to -0.2]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab; Ranked ANCOVA models with covariate adjustment for geographic region and baseline T2 lesion volume was used. Secondary endpoints were analyzed sequentially as: Proportion of participants relapse free at Year 2, Change from baseline in EDSS, Percent change from Baseline in magnetic resonance imaging-T2 hyperintense lesion volume at Year 2, Acquisition of disability measured by multiple sclerosis functional composite. Each endpoint could only be formally tested if prior endpoint was significant; Test type: Superiority or Other; p = 0.3080, Ranked ANCOVA

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 2 years
Description: If a participant experienced both a serious and a non-serious event with the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. The analysis was performed on the safety population, defined as all participants who received any amount of study drug.
Arm/Group | Interferon Beta-1a | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 27/187 | 69/376
Other Adverse Events (participants affected / at risk) | 168/187 | 360/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=187) | Alemtuzumab (N=376)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 2
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 2
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Thyrotoxic crisis (Endocrine disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Meningitis herpes (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Uterine infection (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Thyroxine free increased (Investigations) | 0 | 1
Tri-iodothyronine free increased (Investigations) | 0 | 1
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 13 | 19
Syncope (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Physical assault (Social circumstances) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=187) | Alemtuzumab (N=376)
Anaemia (Blood and lymphatic system disorders) | 11 | 8
Leukopenia (Blood and lymphatic system disorders) | 10 | 11
Lymphopenia (Blood and lymphatic system disorders) | 8 | 26
Neutropenia (Blood and lymphatic system disorders) | 12 | 7
Tachycardia (Cardiac disorders) | 3 | 34
Abdominal pain (Gastrointestinal disorders) | 5 | 21
Abdominal pain upper (Gastrointestinal disorders) | 0 | 22
Diarrhoea (Gastrointestinal disorders) | 6 | 36
Dyspepsia (Gastrointestinal disorders) | 8 | 33
Nausea (Gastrointestinal disorders) | 14 | 65
Vomiting (Gastrointestinal disorders) | 4 | 42
Chest discomfort (General disorders) | 6 | 25
Chills (General disorders) | 3 | 38
Fatigue (General disorders) | 23 | 68
Influenza like illness (General disorders) | 59 | 19
Injection site erythema (General disorders) | 56 | 0
Injection site haematoma (General disorders) | 12 | 1
Injection site pain (General disorders) | 10 | 0
Injection site reaction (General disorders) | 14 | 0
Pain (General disorders) | 5 | 23
Pyrexia (General disorders) | 18 | 138
Bronchitis (Infections and infestations) | 4 | 23
Influenza (Infections and infestations) | 11 | 28
Nasopharyngitis (Infections and infestations) | 25 | 74
Oral herpes (Infections and infestations) | 2 | 40
Rhinitis (Infections and infestations) | 6 | 20
Sinusitis (Infections and infestations) | 9 | 30
Upper respiratory tract infection (Infections and infestations) | 25 | 57
Urinary tract infection (Infections and infestations) | 8 | 64
Contusion (Injury, poisoning and procedural complications) | 11 | 38
Alanine aminotransferase increased (Investigations) | 19 | 2
Aspartate aminotransferase increased (Investigations) | 17 | 3
B-lymphocyte count decreased (Investigations) | 0 | 19
Blood urine present (Investigations) | 6 | 20
CD4 lymphocytes decreased (Investigations) | 4 | 26
CD8 lymphocytes decreased (Investigations) | 5 | 26
T-lymphocyte count decreased (Investigations) | 5 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 48
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 29
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 35
Dizziness (Nervous system disorders) | 8 | 33
Dysgeusia (Nervous system disorders) | 19 | 39
Headache (Nervous system disorders) | 52 | 189
Hypoaesthesia (Nervous system disorders) | 19 | 28
Migraine (Nervous system disorders) | 11 | 15
Multiple sclerosis relapse (Nervous system disorders) | 64 | 65
Paraesthesia (Nervous system disorders) | 13 | 32
Anxiety (Psychiatric disorders) | 10 | 24
Depression (Psychiatric disorders) | 14 | 28
Insomnia (Psychiatric disorders) | 31 | 56
Menorrhagia (Reproductive system and breast disorders) | 2 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 42
Erythema (Skin and subcutaneous tissue disorders) | 6 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 52
Rash (Skin and subcutaneous tissue disorders) | 9 | 174
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 28
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 50
Flushing (Vascular disorders) | 10 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after sponsor published, after a defined period of time after study completion, and/or with written sponsor approval. Generally PI gives sponsor a draft 60 days before publication. Sponsor can ask that confidential information be removed, and can further defer publication upon notifying PI that it will file a patent application on inventions contained in the draft.